CLINICAL TRIAL: NCT04499053
Title: A Phase II Trial of Durvalumab (MEDI4736) and Tremelimumab in Combination With Chemotherapy in HIV-infected Patients With Non-small Cell Lung Cancer
Brief Title: Durvalumab and Tremelimumab in Combination With Chemotherapy in HIV-infected Patients With Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002036
Record Dates: First submitted 2020-07-14; First posted 2020-08-05 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Lung Cancer; Non-Small Cell Lung Cancer; Durvalumab; Tremelimumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- durvalumab (MEDI4736) and tremelimumab (Experimental): Durvalumab in combination with tremelimumab and platinum-based doublet chemotherapy. Only subjects who achieve stable disease or better radiological response after 4 cycles of induction treatment will be eligible to continue study treatment with durvalumab in maintenance.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — durvalumab 1500 mg, intravenous, every 3 weeks for 4 cycles, followed by 1500 mg, intravenous, every 4 weeks (maintenance treatment)
Drug: Tremelimumab — tremelimumab 75 mg, intravenous, every 3 weeks for 4 cycles. A dose of tremelimumab 75 mg will be given at week 16.

SUMMARY:
This is a phase II trial of durvalumab and tremelimumab in combination of platinum-based chemotherapy. Patients with stage IV Non-Small-Cell-Lung Cancer (NSCLC) with human immunodeficiency virus (HIV) infection will be eligible. Patients will receive standard platinum-based chemotherapy plus durvalumab for 4 cycles (every 3 weeks), followed by durvalumab (with or without pemetrexed for non-squamous NSCLC) maintenance therapy. It is hypothesized that Durvalumab and tremelimumab in combination with standard chemotherapy is safe and effective for the treatment of stage IV NSCLC in patients with HIV infection.

DETAILED DESCRIPTION:
This is an open-label, non-randomized phase II trial of durvalumab and tremelimumab in combination with platinum-based doublet chemotherapy. Patients with stage IV NSCLC with HIV infection will be eligible. Patients will receive standard chemotherapy plus durvalumab (1500 mg) and tremelimumab (75 mg) every three weeks for 4 cycles, followed by maintenance treatment with durvalumab (1500 mg Q4W; with or without pemetrexed for non-squamous NSCLC per the discretion of the investigator). A dose of tremelimumab 75 mg will be given at week 16.

Patient will be enrolled into the trial using an optimal two-stage phase II trial design. If 0 of the 7 achieved a response, no further patients will be enrolled in that cohort. If 1 or more of the first 7 patients has a response, accrual would continue until a total of 18 patients have been enrolled in that cohort. Objective response will be evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Safety and tolerability will be evaluated by assessing the incidence of treatment-related grade 3 or higher AEs. Treatment-related grade 3 or higher AEs will be defined as any grade 3 or higher AEs that occur during the first 42 days of treatment and are related to the study treatment. AEs will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

Subjects will receive 4 cycles of combination treatment: durvalumab (1500 mg every 3 weeks) and tremelimumab (75 mg every 3 weeks) in combination with platinum-based doublet chemotherapy. The platinum-based doublet chemotherapies (carboplatin plus paclitaxel/nab-paclitaxel vs. pemetrexed plus carboplatin/cisplatin) are dependent on the tumor histology of the subject (squamous vs. non-squamous). Only subjects who achieve stable disease or better radiological response after 4 cycles of induction treatment will be eligible to continue study treatment in maintenance. The choice to treat non-squamous subjects with pemetrexed maintenance after the 4 induction cycles will be determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage IV NSCLC who had undergone no previous systemic therapy for stage IV disease.
2. Patients with HIV must be on an effective combination anti-retroviral therapy (cART) regimen for ≥ 4 weeks. Also, patients need to meet the following criteria.

   * Documented HIV viral load < 400 copies/mL
   * No AIDS-defining opportunistic infections within the last 12 months
   * No concurrent incurable AIDS-defining malignancy
3. Age > 18 years at time of study entry.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
5. Body weight >30kg
6. Adequate normal organ and marrow function as defined below:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,000 per mm3
   * Platelet count ≥ 100,000 per mm3
   * CD4 T-cell count ≥ 100 per mm3 for HIV-infected patients
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
   * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males: Creatinine CL (mL/min) = [Weight (kg) x (140 - Age)] / [72 x serum creatinine (mg/dL)] Females: Creatinine CL (mL/min) = [Weight (kg) x (140 - Age) x 0.85] / [72 x serum creatinine (mg/dL)]
7. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
8. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
9. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Sensitizing EGFR mutations (deletion in exon 19, L858R in exon 21, G719X, and L861Q) and/or ALK translocations by locally approved laboratory testing including blood-based liquid biopsy.
2. 2. Coinfection of HIV + HBV (coinfection of HIV and HBV allowed if the patient is on appropriate anti-viral therapy for HBV) or HIV + HCV (coinfection of HIV and HCV allowed if HCV is cured or patient is on appropriate anti-viral therapy for hepatitis C). Coinfection of HBV and HCV is allowed if otherwise eligible.
3. No measurable disease.
4. Receipt of the last dose of anticancer therapy (chemotherapy, targeted therapy) ≤ 21 days prior to the first dose of study treatment.
5. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy (chemotherapy, targeted therapy, radiation therapy) with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
6. Patients who have had whole brain radiation therapy (WBRT) during the previous 2 weeks before treatment (no washout period is required for patients who have received stereotactic body radiation therapy).
7. Subject has had major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior to starting study drug or has not recovered from side effects of such procedure (≥ grade 2 AE related to such procedure). Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and subject can be enrolled in the study ≥ 1 week after the procedure.
8. History of allogenic organ transplantation.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   i. Patients with vitiligo or alopecia ii. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement iii. Any chronic skin condition that does not require systemic therapy iv. Patients without active disease in the last 5 years may be included
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
11. Patients with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
12. Previously untreated central nervous system (CNS) metastases or leptomeningeal disease. Patients who have had whole brain radiation therapy (WBRT) during the previous 2 weeks before treatment (no washout period is required for patients who have received stereotactic body radiation therapy).
13. Active tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice).
14. Current or prior use of immunosuppressive medication within 7 days before the first dose of durvalumab. The following are exceptions to this criterion:

    i. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) ii. Systemic corticosteroids at doses not to exceed 20 mg/day of prednisone or its equivalent iii. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) iv. Decreasing dose of systemic corticosteroids after radiation therapy for brain metastasis.
15. Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational product (IP). Note: Patients, if enrolled, should not receive live vaccine whilst receiving study treatment and up to 30 days after the last dose of IP.
16. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control.
17. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
18. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4 within 12 months of the first dose of durvalumab.
19. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | At the end of Cycle 4 (each cycle is 3 weeks)
  Incidence of treatment-emergent Adverse Events according to NCI CTCAE v5.0.
Radiological Response | At the end of Cycle 4 (each cycle is 3 weeks)
  Radiological response will be evaluated using Recist Version 1.1 Criteria

SECONDARY OUTCOMES:
Changes in Viral Load | At the end of Cycle 4 (each cycle is 3 weeks)
  Evaluate changes in viral load with study treatment
Change in Cytokine Secretion Assays | 36 months
  Cytokine secretion assays will be performed on blood samples before, during, and after treatment.
Correlation of Multiplex IHC to response | 36 months
  Baseline immune biomarkers (e.g. PD-L1 expression, composition of T cells in tumor microenvironment) using multiplex IHC will be compared between responders and non-responders to find predictive biomarkers associated with response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chul Kim, MD, Study Chair — Georgetown University
Locations (4):
- United States (4):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Marlene and Stewart Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Harry and Jeannette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No